CLINICAL TRIAL: NCT00505141
Title: Case-Control Study of Urban Environmental Effects on Childhood Leukemia and Brain Cancer
Brief Title: Urban Environmental Exposures and Childhood Cancer
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Other Study IDs: 2004-278
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Brain Cancer; Acute Lymphoblastic Leukemia
Keywords: Childhood Brain Cancer; Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Brain Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The Environmental Protection Agency has recognized that organophosphorus pesticides require close regulation and continued monitoring for human health effects and some (e.g chlorpyrifos) have been phased-out from the consumer market due to the special risk that it posed for children. There is growing evidence in support of the association between pesticide exposure and childhood leukemia. Studies of pesticides and their association with childhood cancer have been limited by study designs, self-reporting and lack of biological measurements. While several large studies in California found little evidence of an association between agricultural pesticide use and childhood leukemia, these results are in contrast with the associations observed with household exposures to pesticides. The real association may depend on timing of exposure, type of pesticide, dose and pathway of exposure. Furthermore, some persons may be more susceptible to the effects of specific pesticides due to inherited mutations in their detoxification pathways.

We are conducting a pilot study to test the hypothesis that environmental exposure to pesticides in pregnancy or during the neonatal period, together with genetic susceptibility may lead to childhood ALL or brain cancer. The study is a multicenter, case-control study, based on collaboration between clinical researchers and basic science research to evaluate the risk for childhood cancer in relation to measured levels of pesticides (and their metabolites) and genetic polymorphisms. Biomarkers will be used to examine the risks of chronic low-dose exposures, and to characterize relationships between specific pesticides, childhood cancer and genetic susceptibility.

Hypothesis: Interaction between environmental factors (pesticides) and maternal or child genetic polymorphisms may lead to childhood cancer.

ELIGIBILITY:
Inclusion Criteria:

* Only newly diagnosed cases of ALL and brain cancers (i.e. diagnosed within the previous 12 months) under the age of 18 years are eligible for this study. These will include live born infants at term or born prematurely, and any cases we are able to ascertain from pediatric hematology records.
* Healthy controls of similar age will be recruited.
* The children must have a parent available to be interviewed who speaks English or Spanish well enough to understand the questionnaire.

Exclusion criteria:

* Subjects with a diagnosis of Down syndrome or other chromosomal disorder, single gene disorder, or recognized multi-organ syndrome will be excluded.
* Non-residents of Maryland, the District of Columbia, and Virginia will be excluded; this will avoid the inclusion of out-of-state case families who traveled a long distance for clinical care, where control sampling would be problematic.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2004-09; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Offie P Soldin, Principal Investigator — Lombardi Comprehensive Cancer Center, Georgetown University Medical Center
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States